CLINICAL TRIAL: NCT01815216
Title: The Effects of Bariatric Surgery on Impulsivity and Attentional Bias to Food Cues
Brief Title: Effect of Gastric Bypass Surgery on Brain Responses
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PH2013b; EPN 2012/451 (Other: Ethical Board Uppsala)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Hormone Responses; Cognitive Health
Keywords: Bariatric surgery; Cognition; Satiety hormones; Brain networks; Inhibitory control; Food intake
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bariatric surgery (Experimental): patients participating in the intervention group , i.e. assessing effects of bariatric surgery on: Brain activity in resting state Memory performance
  Interventions: Procedure: Bariatric surgery; Behavioral: Brain activity in resting state; Behavioral: Memory performance
- Control (Active Comparator): Patients in the control group will not undergo surgery during study.
  These patients will be examined twice:
  1. 9 weeks before the operation (i.e. clinical intervention to reduce body weight has not started).
  2. after 4 weeks of low-calorie diet (which will be a week before their surgery, when patients are in a catabolic metabolism because they eat much less energy than is needed) to assess effect of acute weight loss on: Brain activity in resting state Memory performance
  Interventions: Behavioral: Brain activity in resting state; Behavioral: Memory performance

INTERVENTIONS:
Procedure: Bariatric surgery — Gastric bypass surgery
  Arms: Bariatric surgery
Behavioral: Brain activity in resting state — Measure of activity in brain networks during resting state
Behavioral: Memory performance — Assess concentration in 2D-location task (i.e. "memory game")

SUMMARY:
After obesity surgery gastric bypass (GBP) patients usually lose more than 50% of its former preponderance in relative short time (~ 2 years). But knowledge of the underlying biological mechanisms of decline in body weight is still inadequate.

This project intends to examine patients' background activity in the brain (i.e. "the resting state activity") and brain volume using MRI both before and one year after surgery.

DETAILED DESCRIPTION:
We will also investigate whether hormonal changes in response to food intake after obesity surgery is associated with patients' impulsive control when exposed to pictures of food in the MRI.

ELIGIBILITY:
Inclusion Criteria:

* female
* right-handed
* scheduled for bariatric surgery in the Academic Hospital of Uppsala, Sweden

Exclusion Criteria:

* undergone more than one bariatric surgery
* suffer from mental disorders (depression, phobias, etc.) that can not be controlled with treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in background activity in the brain (resting state activity) after bariatric surgery | 1 year
  Brain's basic activity and structure will be measured on 3 occasions: 4 weeks before bariatric surgery, 4 weeks after surgery and 1 year after surgery, using fMRI.

SECONDARY OUTCOMES:
Change in response inhibition after bariatric surgery | 1 year
  Inhibitory control to food cues will be measured on 3 occasions: 4 weeks before bariatric surgery, 4 weeks after surgery and 1 year after surgery, using a NoGo-Go task.

OTHER OUTCOMES:
Change in memory-function after bariatric surgery ("concentration") | 1 year
  Memory performance will be measured on 3 occasions: 4 weeks before bariatric surgery, 4 weeks after surgery and 1 year after surgery - using a a 2D-object location task ("memory game")

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Sundbom, MD, Study Director — Academic Hospital Uppsala; Christian Benedict, PhD, Study Director — Uppsala University; Pleunie Hogenkamp, PhD, Principal Investigator — Uppsala University
Locations (1):
- Academic Hospital, Uppsala, Sweden